CLINICAL TRIAL: NCT02360852
Title: An Exploratory, Phase IIa Study to Demonstrate the Safety and Efficacy of A4250 in Patients With Primary Biliary Cirrhosis and Cholestatic Pruritus
Brief Title: IBAT Inhibitor A4250 for Cholestatic Pruritus
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: (Expected) side effects
Sponsor: Sahlgrenska University Hospital (Other)
Collaborators: Albireo (Industry)
Responsible Party: Principal Investigator, Hanns-Ulrich Marschall, MD, Sahlgrenska University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A4250 PBC Pruritus
Record Dates: First submitted 2015-01-14; First posted 2015-02-11 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Biliary Cirrhosis, Primary
MeSH Terms: conditions — Liver Cirrhosis, Biliary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A4250 (Experimental): A4250 once daily
  Interventions: Drug: A4250

INTERVENTIONS:
Drug: A4250 — A4250 once daily
  Other Names: IBAT Inhibitor A4250

SUMMARY:
This study will evaluate the safety, tolerability and influence on itching, bile acids and liver enzyme changes in patients with PBC (Primary Biliary Cirrhosis) treated with A4250

DETAILED DESCRIPTION:
A4250PBCpruritus (EudraCT 2014-004070-42) is an open-label exploratory study.

The primary objective of this study is to assess the safety and tolerability of A4250, 1.5 - 3 mg orally during a four-week treatment period, in patients with PBC and cholestatic pruritus, as determined by the occurrence of treatment-emergent serious adverse events (SAEs).

Other safety objectives of this study include assessment of the safety and tolerability of A4250 during a four-week treatment period, as determined by the occurrence of treatment-emergent adverse events (AEs) and changes in other safety parameters including liver and kidney function tests and vital signs.

Exploratory efficacy objectives of this study are to demonstrate the efficacy of A4250 orally on pruritus variables and on QoL and lysophosphatidic acid formation as well as evaluation of changes in pharmacodynamic parameters of bile acid metabolism such as serum and fecal bile acids, C4 and fibroblast growth factor 19 (FGF19) assessments and assessment of surrogate markers of cholestatic liver disease such as alkaline phosphatase, transaminases and bilirubin.

ELIGIBILITY:
Major Inclusion Criteria:

* Diagnosis of PBC or PBC-Autoimmune hepatitis overlap as established according to American Association for the Study of Liver Diseases/European Association for the Study of Liver (AASLD/EASL) definitions. Definite or probable PBC diagnosis, as demonstrated by the presence of ≥ 2 of the following 3 diagnostic factors:
* History of elevated alkaline phosphatase (ALP) levels (>1.67 ULN) for at least 6 months prior to Day 1
* Positive antimitochondrial antibodies (AMA) titer or if AMA negative or in low titer (<1:80) PBC specific antibodies (anti-GP210 and/or anti-SP100 and/or antibodies against the major M2 components (PDC-E2, 2-oxo-glutaric acid dehydrogenase complex)
* Liver biopsy consistent with PBC;
* Ursodeoxycholic acid (UDCA) non-responders defined as >6 months of UDCA and at the time of enrolment a serum ALP >1.67 ULN;
* Laboratory markers of cholestasis identified within 3 months of Visit 1;
* Treatment with cholestyramine at a dose >4g BID or colestipol > 5mg for at least 3 months;
* The patient has a VAS-Itch of at least 30 mm during the day before baseline (Visit 2);
* The patient is a male or non-pregnant female ≥18 years of age and ≤80 years of age with body mass index (BMI) ≥18.5 but <35 kg/m2;

Major Exclusion Criteria:

* Any condition that, in the opinion of the Investigator constitutes a risk for the patient or a contraindication for participation and completion of the study, or could interfere with study objectives, conduct, or evaluations;
* Jaundice of extrahepatic origin;
* The patient has a structural abnormality of the GI tract;
* The patient has a known, active, clinically significant acute or chronic infection, or any major episode of infection requiring hospitalization or treatment with parenteral anti infectives within 4 weeks of treatment start (study day 1) or completion of oral anti-infective treatment within 2 weeks prior to start of screening period;
* The patient has unexplained and clinically significant GI alarm signals (e.g., lower GI bleeding or heme-positive stool, iron-deficiency anaemia, unexplained weight loss) or systemic signs of infection or colitis;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2015-01; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
•Safety and Tolerability assessed by the occurrence of treatment-emergent SAEs during the four weeks of treatment with A4250 | 4 weeks

SECONDARY OUTCOMES:
Safety laboratory measurements | 4 weeks
  Changes in safety laboratory test results (including hematology, clinical chemistry and urinalysis) from baseline to Day 28 of A4250 treatment
VAS-Itch | 4 weeks
  Change in VAS-Itch (most severe itch during last 24 hrs) during the fourth treatment week of A4250
Itching scale | Four weeks
  Change in PBC40
Bile acid evaluation | Four weeks
  Change in serum and fecal bile acids (BAs)
Liver biochemistry | Four weeks
  Change in ALP

CONTACTS AND LOCATIONS:
Overall Officials: Hanns-Ulrich Marschall, MD, Principal Investigator — Sahlgrenska Academy, Institute of Medicine,
Locations (1):
- Sahlgrenska Academy, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No